CLINICAL TRIAL: NCT01911039
Title: A Phase 1 Safety and Tolerability Study of Infused Donor T Regulatory Cells in Steroid Dependent/Refractory Chronic Graft Versus Host Disease
Brief Title: Phase 1 Infused Donor T Regulatory Cells in Steroid Dependent/Refractory Chronic GVHD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laura Johnston (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Laura Johnston, Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-27285; BMT253 (Other: OnCore)
Record Dates: First submitted 2013-07-15; First posted 2013-07-30 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Graft Versus Host Disease; Allogeneic Hematopoietic Cell Transplant Recipient
Keywords: GVHD; cGVHD
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Regulatory T Cells (Experimental): Cohort 1 at 1x105 Treg cells/kg, Cohort 2 at 5x105 Treg cells/kg and Cohort 3 at 1.5x106 Treg cells/kg with an extension phase at the MTD (or maximum administered dose if the MTD is not reached).
  Interventions: Biological: Regulatory T Cells

INTERVENTIONS:
Biological: Regulatory T Cells
  Other Names: donor Treg cell

SUMMARY:
Chronic graft versus host disease (cGVHD) is a common complication of bone marrow or hematopoietic cell transplant from another person (allogeneic transplant). This study will determine if subjects with steroid dependent/refractory cGVHD can tolerate infusion of donor regulatory T cells and whether their cGVHD responds to the infusion.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Determine the safety and tolerability of donor T regulatory (Treg) cell infusions in subjects with steroid dependent/refractory chronic graft versus host disease.

SECONDARY OBJECTIVES:

1. Determine the quantitative blood Treg cell changes following the cell infusions
2. Determine clinical efficacy of donor Treg cells as failure-free survival (FFS) defined by the absence of a new immunosuppressive therapy added, non-relapse mortality, and recurrent malignancy at Day 180 after the first Treg infusion
3. In addition to FFS, the study will measure the change in:

   1. cGVHD symptom burden measured by the Lee cGVHD Symptom Scale by increase in >7 points
   2. NIH organ-specific cGVHD scale
   3. The reduction in daily corticosteroid requirement of prednisone to <=0.25 mg/kg-day at Day 180 after the first Treg infusion

ELIGIBILITY:
Inclusion Criteria:

* Steroid dependent/refractory cGVHD defined as:

  * Steroid dependent disease: Persistent cGVHD manifestations requiring a glucocorticoid dose >= prednisone 0.25 mg/kg/day (0.5 mg/kg orally [po] every other day) for at least 12 weeks
  * Steroid refractory disease: Progressive cGVHD manifestations despite treatment with a glucocorticoid dose >= prednisone 0.5 mg/kg/day (1 mg/kg po every other day) for at least 4 weeks
* Participants must be receiving systemic glucocorticoid therapy for cGVHD; all immunosuppressive therapy may include but not be limited to tacrolimus, sirolimus, CellCept, cyclosporine, and systemic corticosteroid must be at stable doses for 28 days prior to the first cell infusion
* Chronic GVHD manifestations that can be followed on physical or laboratory exam; these include but are not necessarily limited to:

  * Skin changes
  * Oral mucosa changes
  * Bronchiolitis obliterans
  * Ocular changes
* Karnofsky performance status >= 60
* Serum creatinine =< 2 mg/dL
* Absolute neutrophil count (ANC) > 1 x 10^9/L
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 20 x upper limit of normal (ULN) or
* Total bilirubin =< 10 x ULN
* Allogeneic hematopoietic cell transplant recipient
* Transfusion independent
* Oxygen saturation during exertion is maintained at >= 88% on room air
* Does not have clinically significant, symptomatic uncontrolled heart disease (e.g., unstable angina, congestive heart failure, or uncontrolled hypertension)
* DONOR: Age >= 18 to =< 75 years old
* DONOR: Karnofsky performance status of >= 70% defined by institutional standards
* DONOR: Must be the same sibling donor from whom the recipient's blood and marrow graft was collected for the original allogeneic transplant that is human leukocyte antigen (HLA) 7/8 or 8/8 matched at the HLA-A, B,C, DRB1
* DONOR: Serologies for human immunodeficiency virus (HIV) antigen (Ag), HIV 1 and HIV 2 antibody (Ab), human T-lymphotropic virus type I (HTLV 1) and HTLV 2 Ab, hepatitis B surface antigen (sAg) or polymerase chain reaction positive (PCR+), or hepatitis C Ab or PCR+, Syphilis (Treponema) screen and HIV 1 and hepatitis C by nucleic acid testing (NAT) have been collected prior to apheresis
* DONOR: Female donors of child-bearing potential must have a negative serum or urine beta-human chorionic gonadotropin (HCG) test within three weeks of apheresis
* DONOR: Capable of undergoing leukapheresis, have adequate venous access, and be willing to undergo insertion of a central catheter should leukapheresis via peripheral vein be inadequate
* DONOR: Donor selection will be in compliance with 21 Code of Federal Regulations (CFR) 1271

Exclusion Criteria:

* Original transplant utilized an unrelated donor graft
* Uncontrolled infections that are not responsive to antimicrobial therapy
* Progressive malignant disease, including post-transplant lymphoproliferative disease unresponsive to therapy
* Second malignancy except for skin cancer within the last 5 years
* Received any investigational agent =< 28 days before Treg infusions
* Received filgrastim (GCSF) treatment within one month of enrollment
* Received a donor lymphocyte infusion (DLI) or hematopoietic cell transplantation (HCT) within 3 months of enrollment
* DONOR: Evidence of active infection or viral hepatitis
* DONOR: HIV positive
* DONOR: Pregnant donor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-07; Primary Completion 2017-12-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
The frequency of adverse events related to the donor Treg infusions (e.g., grade III-IV aGVHD by the modified Keystone criteria and grade 3 or higher infusional toxicities graded according to the CTCAE v. 4) | Up to day 180
  For infusion-related toxicities, recipients will be monitored for 1 hour after the Treg infusion. Additional toxicities which may occur during the first 28 days after the Treg infusions will count towards the assessment of safety and tolerability (DLT assessment) (e.g., development of aGVHD). Acute GVHD will be assessed using the modified Keystone criteria on Days 14, 28, 42, 56, 84 and 180 after the Treg infusion (or if the subject is exhibiting signs of aGVHD in-between study visits). Dose limiting toxicities are defined in Section 8. Only toxicities which occur during the first 28 days after the cell infusion will count towards the assessment of DLTs. A dose of Treg will be considered safe if DLTs occur in only 1/6 or 0/3 members of the cohort during the dose-escalation phase.

SECONDARY OUTCOMES:
Change in absolute blood Treg levels | Baseline to day 42
  The change in Treg cell counts from baseline to post infusion will be depicted in boxplots of both relative proportion and absolute numbers. Mean log (fold change) and confidence intervals will be calculated.
Improvement in Failure Free Survival (FFS) over cGVHD | At day 180
  FFS is defined as the absence of a third line therapy (treatment failure). Estimated by the Kaplan-Meier product-limit method, with standard confidence limits.
Successful achievement of cGVHD partial response or Complete response by the NIH consensus criteria | Up to day 180
  1. Complete Response (CR) - Complete resolution of all reversible manifestations of cGVHD. Irreversible manifestations will be defined as (NIH consensus criteria) are: ocular xerosis, esophageal stricture, and bronchiolitis obliterans.
  2. Partial Response (PR) - At least a 25% absolute or 50% relative change (whichever is greater) when comparing start and end measurements in one cGVHD manifestation without worsening in the other manifestations.
  The results will be summarized in tabular form, with confidence intervals for the trinomial proportions.
The ability to reduce steroid requirements to <0.25 mg/kg-day | At day 180
Change in >7 points on the Lee cGVHD Symptom scale relates to improvement in quality of life | Baseline to day 180
  A one-sample t-test will be used on the change in scale from baseline to months 1, 3, and 6.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Johnston, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States